CLINICAL TRIAL: NCT03226223
Title: Using Pharmacogenetics to Better Evaluate Naltrexone for Treating Stimulant Abuse
Brief Title: Pharmacogenetics of Naltrexone for Stimulant Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jermaine Jones, Assistant Professor of Clinical Neurobiology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: #7347
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Substance Use Disorders; Methamphetamine Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will complete two testing sessions in which the effects of oral naltrexone (0 mg & 50 mg) will be tested in combination with intranasal methamphetamine. Participants will complete two testing sessions (naltrexone 0 mg + Methamphetamine & naltrexone 50 mg + methamphetamine), in randomized order.
Who Masked: Participant
Masking Description: Participants and study staff conducting the lab sessions will be blinded to the treatment condition (i.e., naltrexone 0 mg or 50 mg)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naltrexone 0 mg (Placebo Comparator): This aim assess the effects of pretreatment with 0 mg of naltrexone on laboratory measures of the abuse potential of methamphetamine (30mg/70 kg).
  Interventions: Drug: Intranasal Methamphetamine
- Naltrexone 50 mg (Experimental): This aim assess the effects of pretreatment with 50 mg of naltrexone on laboratory measures of the abuse potential of methamphetamine (30mg/70 kg).
  Interventions: Drug: Intranasal Methamphetamine

INTERVENTIONS:
Drug: Intranasal Methamphetamine — Intranasal Methamphetamine HCL administered at a dose of 30mg per 70 kg of the participants' body weight)

SUMMARY:
This investigation will be the first study assessing genetic modulation of naltrexone's NTX effects upon the abuse liability of a stimulant drug (methamphetamine). The study team will assess the ability of oral NTX to block the reinforcing and positive subjective effects of intranasal (IN) methamphetamine (30mg/70kg). This investigation could identify an important Gene x Pharmacological interaction, contributing to the personalization of stimulant abuse pharmacotherapy.

DETAILED DESCRIPTION:
A recent meta-analysis concluded that the OPRM1 A118G SNP (rs1799971) significantly moderates the treatment efficacy of Naltrexone (NTX) in treating alcohol abuse, increasing the treatment efficacy by over 2-fold among G-allele carriers (AG/GG). The proposed application would be the first to investigate the moderating effect of this genotype in the efficacy of NTX to treat stimulant abuse. More specifically, the study team proposes to investigate the interaction between NTX and intranasal (IN) methamphetamine (30mg/70kg). Participants who meet DSM criteria for mild-to-severe stimulant use disorder (N=up to 70) will complete 4 testing sessions where drug effects are tested following pretreatment with NTX (0, 50 mg). Naltrexone pretreatment effects upon the abuse liability of IN methamphetamine will be assessed using self-report measurements of positive subjective effects and drug self-administration. Medication effects on these validated predictors of abuse potential will be compared between A118G A allele homozygotes (AA) and G-allele carriers (AG/GG; an anticipated 25% of the total sample), in order to assess genetic moderation of treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 21 to 50 years
2. DSM-5 criteria for mild-to-severe stimulant use disorder, along with intravenous, intranasal or smoked use of amphetamine-type stimulants in amounts equal to or greater than administered in the current study.
3. Able to give written informed consent to participate.
4. Females must be either post-menopausal, surgically sterilized, or using an acceptable method of contraception (double-barrier method like a condom with a spermicidal lubricant) to participate in this study.
5. Racially Caucasian or of European descent.

Exclusion Criteria:

1. Currently seeking treatment for a substance use disorder.
2. DSM-5 criteria for moderate-to-severe substance use disorders (except those involving cocaine, amphetamines and nicotine).
3. Psychiatric condition that may affect the participants' ability to provide informed consent (e.g., psychotic disorder), or make participation hazardous for the participant or study staff (e.g., severe depression/suicidality, or risk of violence).
4. Uncontrolled neurological, cardiovascular, and hepatic diseases, active tuberculosis, or any other disorder that might make administration of study medications hazardous.
5. Gastrointestinal or renal disease that would significantly impair absorption, metabolism or excretion of study drug, or require medication or medical treatment.
6. Current treatment with a psychotropic medication that in the physician's judgement would interfere with the study endpoints.
7. History of allergy, adverse reaction, or sensitivity to amphetamines.
8. Medical conditions that may make study participation hazardous:

   * History of seizures or cardiac risk conditions (unstable angina, cardiac arrhythmias, chest pain, strong palpitations (subjectively defined as the feeling that the heart is beating too hard, too fast, skipping a beat, or fluttering).
   * Elevated liver function tests (i.e., AST and ALT > 3 times the upper limit of normal).
   * Impaired renal function (creatinine > 1.2).
   * Hypertension (>140/90).
   * Asthmatic symptoms within the past 3 years.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jermaine Jones, PhD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone 0mg First, Then Naltrexone 50mg: This aim assess the effects of pretreatment with 0 mg of naltrexone on laboratory measures of the abuse potential of methamphetamine (30mg/70 kg).
  Intranasal Methamphetamine: Intranasal Methamphetamine HCL administered at a dose of 30mg per 70 kg of the participants' body weight)
- Naltrexone 50mg First, Then Naltrexone 0mg: This aim assess the effects of pretreatment with 50 mg of naltrexone on laboratory measures of the abuse potential of methamphetamine (30mg/70 kg).
  Intranasal Methamphetamine: Intranasal Methamphetamine HCL administered at a dose of 30mg per 70 kg of the participants' body weight)
Period: Overall Study
Arm/Group | Naltrexone 0mg First, Then Naltrexone 50mg | Naltrexone 50mg First, Then Naltrexone 0mg
Started | 10 | 8
Completed | 8 | 6
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data are provided for participants who completed both conditions N=14.
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone 0mg First, Then Naltrexone 50mg | Naltrexone 50mg First, Then Naltrexone 0mg | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (6.5) | 31.7 (9.3) | 33.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Self-Administration
Description: To assess the reinforcing effects of methamphetamine, participants complete a drug self-administration procedure. The outcome measure for this procedure is the number of operant responses (clicks on a mouse) participant are willing to make in order to receive drug (methamphetamine).
Time Frame: 1 day.
Measure: Mean (Standard Deviation); unit: Clicks on a computer mouse
Arm/Group | Naltrexone 0 mg | Naltrexone 50 mg
Number analyzed (Participants) | 14 | 14
Clicks on a computer mouse | 8890 (3509) | 7116 (3080)

2. Secondary Outcome: Positive Subjective Effects of Methamphetamine.
Description: Participant ratings of methamphetamine "Liking," on a 100 mm visual analog scale. Participants are asked to indicate on a 100 mm line the extent to which they agree with the description of the drug provided. The 0 mm end of the line indicates "Not at All," while the 100 mm indicates "Extremely."
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone 0 mg | Naltrexone 50 mg
Number analyzed (Participants) | 14 | 14
units on a scale | 53.6 (38.9) | 57.2 (32.5)

ADVERSE EVENTS:
Time Frame: 1 Month
Arm/Group | Naltrexone 0 mg | Naltrexone 50 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03226223/Prot_SAP_000.pdf